CLINICAL TRIAL: NCT03030755
Title: Corneal Elastography and Patient Specific Modeling
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, William Dupps Jr., MD, Staff Physician, The Cleveland Clinic
Other Study IDs: 13-213
Record Dates: First submitted 2017-01-11; First posted 2017-01-25 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-09

CONDITIONS: Cornea; Ectasia; Refractive Errors; Keratoconus
MeSH Terms: conditions — Corneal Diseases; Dilatation, Pathologic; Refractive Errors; Keratoconus | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Optical coherence tomography

SUMMARY:
The goal of this research is to develop measurement tools and simulation technology for characterizing and predicting individual responses to corneal treatments and for advancing understanding of corneal ectasia risk factors. Patients who either 1) have keratoconus and are being evaluated for corneal crosslinking or 2) have refractive error and are being evaluated for refractive surgery procedures such as LASIK will have their eyes imaged to assess their mechanical properties and will have computational simulations performed to predict the response to treatment. One aim of the study is to test the hypothesis that computational models can predict the cornea's shape changes within clinically acceptable limits of error.

DETAILED DESCRIPTION:
The mechanical condition of the cornea is an important but elusive property of the eye to characterize. Weakness in the cornea is thought to be one of the primary causes of corneal ectasia, a major cause of visual impairment worldwide. Corneal weakness is also important to identify in refractive surgery candidates since such surgeries often involve tissue removal that could lead to corneal instability in certain predisposed patients.

In this study, subjects will undergo imaging with an optical coherence tomography (OCT)-based system to characterize corneal biomechanical properties. In addition, computational representations of the eye will be built from images and interventions will be simulated and compared to actual treatment outcomes. No investigational procedures or study-specific interventions other than imaging are involved.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with keratoconus diagnosed by standard criteria, including topographic steepness, irregular astigmatism with a pattern consistent with keratoconus.
* Any patient deemed a candidate for LASIK (laser vision correction) and scheduled for surgery.

Exclusion Criteria:

* Inability to provide informed consent, including non-English speaking (if interpreter not available) and cognitively/mentally impaired (if legal guardian not available).

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with refractive error who present for screening for refractive surgery and individuals with keratoconus who are evaluatedat the Cole Eye Institute in Cleveland, Ohio
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Predictive accuracy of computational models in corneal surgery | 3 month
  Computational model predictions of corneal interventions will be compared to actual clinical outcomes for each enrolled subject

CONTACTS AND LOCATIONS:
Overall Officials: William Dupps, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation Cole Eye Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ford MR, Dupps WJ Jr, Rollins AM, Sinha RA, Hu Z. Method for optical coherence elastography of the cornea. J Biomed Opt. 2011 Jan-Feb;16(1):016005. doi: 10.1117/1.3526701. PMID 21280911
- [Background] Sinha Roy A, Dupps WJ Jr. Patient-specific computational modeling of keratoconus progression and differential responses to collagen cross-linking. Invest Ophthalmol Vis Sci. 2011 Nov 25;52(12):9174-87. doi: 10.1167/iovs.11-7395. PMID 22039252